CLINICAL TRIAL: NCT05140044
Title: Longitudinal Home-based Evaluation of Balance and Exercise in Older Adults With and Without a History of Falls
Brief Title: Use of a Smartphone to Assess Balance and Provide Intervention to Older Adults at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Binghamton University (Other)
Responsible Party: Principal Investigator, Vipul Lugade, Associate Professor and Director of Motion Analysis Research Laboratory, Binghamton University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: Smartphone Balance & Exercise
Record Dates: First submitted 2021-11-09; First posted 2021-12-01 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fall
Keywords: Older Adults; Balance; Smartphone; Home-based Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home - Paper Intervention (Active Comparator): Older adults who are given a 4-week paper-based balance intervention program. Performed 3days/week for 30min/day over the course of a 4-week period using printed materials with text instruction and images.
  Interventions: Other: Balance Exercises - Traditional Paper Delivery
- Home - Smartphone Intervention (Experimental): Older adults who are given a 4-week home-based balance exercise program. Performed 3days/week for 30min/day over the course of a 4-week period using participants' smartphones.
  Interventions: Device: Balance Exercises - Smartphone Delivery

INTERVENTIONS:
Device: Balance Exercises - Smartphone Delivery — 1st week: standing balance tasks; 2nd week: standing with arm manipulation tasks; 3rd week: gait balance tasks; 4th week: gait with arm manipulation tasks.
  Arms: Home - Smartphone Intervention
Other: Balance Exercises - Traditional Paper Delivery — 1st week: standing balance tasks; 2nd week: standing with arm manipulation tasks; 3rd week: gait balance tasks; 4th week: gait with arm manipulation tasks.
  Arms: Home - Paper Intervention

SUMMARY:
Approximately one-third of older adults report one or more falls each year, with devastating physical, psychological, social, and financial consequences. Conventional gait analysis performed in a controlled laboratory environment can identify balance deficits, but unfortunately, such tools are bulky, time-consuming, and dependent on qualified technicians to properly collect and evaluate the data. Furthermore, these one-time gait and balance assessments cannot monitor changes in ambulatory strategies longitudinally and do not reflect performance in real-life environments, where falls commonly occur. While recent developments in smartphone-based evaluations have demonstrated great utility and accuracy in assessing gait performance, it is vital to evaluate participant compliance, ease-of-use, and feasibility of this technology using a smartphone in the home environment.

It is also paramount that interventions which improve balance be accessible to older adults. While four-week balance training routines have been shown to improve balance performance among older adults, it is unknown whether such interventions can be conducted remotely in a safe and compliant manner. Furthermore, the retention of balance function following intervention is unclear. Subsequently, the goals of this study are to evaluate technology that can both remotely monitor balance and prescribe intervention to older adults. With the current burdens on the health care system and the burgeoning population of older adults, it is essential that tools be provided to older adults that are easy to follow, attractive, and improve balance performance.

Therefore, the objective of this project is to investigate the utility of a valid, easily accessible, smartphone application to assess balance and provide personalized exercise for older adults as a stand-alone, field-based medical device. The aims of this proposal are to (1) utilize a smartphone application to longitudinally evaluate gait and standing balance over an 8-week period in the home environment among 30; and (2) determine the feasibility and efficacy of a smartphone application to promote exercise and evaluate gait changes for up to 2 months in this older adult population following a 4-week balance intervention. The long-term goal of this project is to provide a holistic home-based gait monitoring and intervention tool for integration in routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Able to ambulate at least 10 meters without an assistive device.
* Cognitively intact based on scoring 18/22 or greater on the Montreal Cognitive Assessment (MOCA) - Blind.

Exclusion Criteria:

* Lower limb amputation
* Lower limb arthroplasty
* Visual impairment uncorrectable with lenses
* Uncontrolled hypertension or diabetes
* Neurological or musculoskeletal impairment
* Persistent symptoms of dizziness or lightheadedness

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Dual Task Gait Velocity | Baseline
  self-selected walking speed under dual task gait/cognitive conditions
Dual Task Gait Velocity | One-month following baseline
  self-selected walking speed under dual task gait/cognitive conditions
Dual Task Gait Velocity | Two-months following baseline
  self-selected walking speed under dual task gait/cognitive conditions

SECONDARY OUTCOMES:
Dual Task Verbal Reaction Time | Baseline
  Time taken to verbally respond to auditory stimulus under dual task gait/cognitive conditions
Dual Task Verbal Reaction Time | One-month following baseline
  Time taken to verbally respond to auditory stimulus under dual task gait/cognitive conditions
Dual Task Verbal Reaction Time | Two-months following baseline
  Time taken to verbally respond to auditory stimulus under dual task gait/cognitive conditions
Dual Task Standing Balance | Baseline
  Path of Center of Pressure (COP) during standing and performing secondary cognitive task
Dual Task Standing Balance | One-month following baseline
  Path of COP during standing and performing secondary cognitive task
Dual Task Standing Balance | Two-months following baseline
  Path of COP during standing and performing secondary cognitive task

OTHER OUTCOMES:
Single Task Gait Velocity | Baseline
  Level walking speed
Single Task Gait Velocity | One-month post baseline
  Level walking speed
Single Task Gait Velocity | Two-months post baseline
  Level walking speed
Singe Task Reaction Time | Baseline
  Time taken to verbally respond to auditory stimulus while sitting
Singe Task Reaction Time | One-month post baseline
  Time taken to verbally respond to auditory stimulus while sitting
Singe Task Reaction Time | Two-months post baseline
  Time taken to verbally respond to auditory stimulus while sitting

CONTACTS AND LOCATIONS:
Locations (1):
- Binghamton University - Motion Analysis Laboratory, Binghamton, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) including demographic, gait, posture, and cognitive results as well as exercise conditions will be shared.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication.
Access Criteria: IPD will be shared with other researchers on a case by case basis.